CLINICAL TRIAL: NCT05121571
Title: The Efficacy and Safety of Retreatment With Hepatic Arterial Infusion Chemotherapy With Oxaliplatin, Fluorouracil, and Leucovorin vs Sorafenib for Patients Who Showed Transarterial Chemoembolization-resistant: a Retrospective Study
Brief Title: The Efficacy and Safety of HAIC With FOLFOX vs Sorafenib for Patients Who Showed TACE-resistant: a Retrospective Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Shi Ming, Proffessor, Sun Yat-sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SH-4
Record Dates: First submitted 2021-11-14; First posted 2021-11-16 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-11

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; TACE failure; Sorafenib; Hepatic arterial infusion chemotherapy; Oxaliplatin, fluorouracil, and leucovorin
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HAIC of FOLFOX (Experimental): Retreatment With hepatic arterial infusion chemotherapy of oxaliplatin , fluorouracil, and leucovorin
  Interventions: Procedure: HAIC
- Sorafenib (Active Comparator)
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Procedure: HAIC — administration of Oxaliplatin , fluorouracil, and leucovorin via the tumor feeding arteries
  Arms: HAIC of FOLFOX
Drug: Sorafenib — sorafenib 400mg bid
  Arms: Sorafenib

SUMMARY:
Transarterial chemoembolization (TACE) is considered the gold standard for treating intermediate-stage hepatocellular carcinoma (HCC). However, any treatment guidelines do not specify the criteria for repeating TACE. This study was to compare HAIC with FOLFOX with sorafenib who showed TACE-resistant.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with HCC according to the European Association for the Study of the Liver (EASL) diagnostic criteria
* TACE failure/refractoriness by Liver Cancer Study Group of Japan (LCSGJ) criteria
* Without extrahepatic metastasis
* The following laboratory parameters:

Platelet count ≥ 60,000/μL Hemoglobin ≥ 8.5 g/dL Total bilirubin ≤ 1.5 mg/dL Serum albumin ≥ 35 g/L ASL and AST ≤ 5 x upper limit of normal Serum creatinine ≤ 1.5 x upper limit of normal INR ≤ 1.5 or PT/APTT within normal limits Absolute neutrophil count (ANC) >1,500/mm3

Exclusion Criteria:

* Known history of HIV
* History of organ allograft
* Patients with clinically significant gastrointestinal bleeding within 30 days prior to study entry.
* Serious non-healing wound, ulcer, or bone fracture
* Evidence of bleeding diathesis.
* Any other hemorrhage/bleeding event > CTCAE Grade 3 within 4 weeks of first dose of study drug

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2016-04-21 (Actual); Primary Completion 2018-12-12 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Progression free survival | 12 months

SECONDARY OUTCOMES:
Number of Adverse Events | 30 days
overall survival | 24 months
tumor response | 6 months
  RECIST 1.1

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Center Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Huang Y, Zhang L, He M, Lai Z, Bu X, Wen D, Li Q, Xu L, Wei W, Zhang Y, Zhou Z, Chen M, Guo R, Shi M, Kan A. Hepatic Arterial Infusion of Oxaliplatin, Fluorouracil, and Leucovorin Versus Sorafenib for Hepatocellular Carcinoma Refractory to Transarterial Chemoembolization: Retrospective Subgroup Analysis of 2 Prospective Trials. Technol Cancer Res Treat. 2022 Jan-Dec;21:15330338221117389. doi: 10.1177/15330338221117389. PMID 36529949